CLINICAL TRIAL: NCT03987425
Title: Effect of the Intervention With Continuous Positive Pressure (CPAP) on Nocturnal Blood Pressure (BP) in Normotensive Patients With Nondipper Circadian Pattern and Sleep Apnea-hypopnea Syndrome (SAHS)
Brief Title: Normotensive OSA Patients With Nondipper Circadian Blood Pressure Pattern
Acronym: Nondipper-OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Collaborators: Societat Catalana de Pneumologia (Unknown)
Responsible Party: Principal Investigator, Ferran Barbe, Medical Doctor, Chair Respiratory Medicine, Sociedad Española de Neumología y Cirugía Torácica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nondipper-OSA
Record Dates: First submitted 2019-06-10; First posted 2019-06-17 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Normotensive; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP treatment (Experimental): Group of patients who will receive CPAP treatment
  Interventions: Device: CPAP treatment
- Conservative measures (No Intervention): Group of patients who will receive conservative treatment based on hygienic-dietetic measures

INTERVENTIONS:
Device: CPAP treatment — In this group of patients (CPAP group) will be prescribed CPAP treatment at optimal pressure. It will be performed a CPAP titration with an automatic or manual CPAP according to usual clinical practice.
  Arms: CPAP treatment

SUMMARY:
The principal objective is to evaluate the effect of CPAP treatment on blood pressure (BP) in normotensive patients with nondipper circadian pattern with sleep apnea-hypopnea syndrome (SAHS). The secondary objectives are: i) To evaluate the prevalence of the different circadian patterns of BP in ambulatory blood pressure monitoring (ABPM) ii) To establish the relationship between CPAP compliance and BP response; iii) Identify which ABPM variables and biomarkers are related to BP response; iv) Evaluate changes in the biomarkers' profile after CPAP treatment.

Methodology: Open-label, parallel, prospective, randomized and controlled trial including normotensive patients with nondipper circadian pattern diagnosed with severe SAHS without significant somnolence. 64 patients with nondipper circadian pattern will be included and will be randomized to receive CPAP (32) or conservative treatment (32). ABPM and blood sample collection will be performed at the beginning of the study and at 3 months.

DETAILED DESCRIPTION:
1. Recruitment: Normotensive subjects referred to the sleep unit of the Hospital Santa Maria (Spain) who are diagnosed of severe OSA (AHI≥30) by a sleep study and nondipper circadian blood pattern confirmed by ABPM and who do not present significant somnolence (Epworth≤18) will be included in the study.
2. Definition of the groups: Patients will be randomized to receive one of the following treatments:

   * CPAP: Patients who will receive CPAP treatment. The CPAP titration will be carried out with an automatic or manual CPAP according to usual clinical practice.
   * Conservative treatment: Patients who will receive conservative treatment based on hygienic-dietetic measures.
3. Randomization: It will be carried out with an automated platform
4. Duration of the treatment: All patients randomized to CPAP will begin the treatment as soon as possible after randomization, and will continue treatment until the study ends (3 months).

   Patients who interrupt treatment will be excluded from the study. ABPM and blood sample collection will be performed on all included patients at the beginning of the study and at 3 months under treatment (CPAP or conservative care).
5. Follow-up: All patients will be evaluated at the beginning of the study (T0), at first month (T1) and at three months (T2), during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years of age
* Referred to the sleep unit for suspected OSA
* Being normotensive and presenting an AHI ≥ 30 in the sleep study
* Signature of the informed consent.

Exclusion Criteria:

* Previous CPAP treatment
* Significant somnolence defined by an Epworth Sleepiness Scale (ESS) score higher than 18
* Psychophysical inability to complete questionnaires
* Previous diagnosis or suspicion of another sleep disorder
* Presence of more than 50% of central apneas or Cheyne-Stokes respiration
* Having a serious chronic disease: neoplasia, renal failure, severe chronic obstructive pulmonary disease, chronic depression and other chronic limiting diseases
* Medical history that may interfere with the objectives of the study or, in the opinion of the researcher, may compromise the conclusions
* Any medical, social or geographical factor that may endanger the patient's compliance
* Having a profession of high risk (professional driver).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Effect of CPAP treatment on BP in normotensive nondipper patients with severe OSA | 3 years
  Change in mmHg in blood pressure monitoring parameters after 3 months of treatment

SECONDARY OUTCOMES:
Prevalence of the different circadian BP patterns (dipper /nondipper) in the ABPM of normotensive subjects diagnosed with severe OSA without significant somnolence (Epworth≤18) | 3 years
  The prevalence of each circadian patterns will be calculated from the baseline ambulatory blood pressure monitoring data
Relationship between compliance with CPAP treatment and the blood pressure change in normotensive nondipper patients with OSA | 3 years
  The relation between CPAP compliance (mean hours per night) and change in mean nighttime BP using multivariate models in patients randomized to CPAP treatment.
Identify predictors of nocturnal blood pressure response to CPAP treatment | 3 years
  Among all the variables recorded in the 24h-ambulatory blood pressure monitoring (different to circadian blood pressure) the investigators will proceed to the identification of variables that are related to the change in mean nocturnal BP in normotensive nondipper-OSA patients treated with CPAP.
Changes in the biomarkers' profile (miRNAs) in normotensive nondipper-OSA patients after CPAP treatment | 3 years
  The miRNAs profile will be evaluated at baseline and after 3 months of CPAP treatment in order to evaluate changes related to CPAP treatment.
  Learning Phase: complete profile analysis (754 miRNAs) will be carried out in 24 patients representative of the change in BP in treated patients. The miRNAs associated with the change in BP will be identified from the 754 miRNAs potentially present in serum and plasma.
  Validation Phase: Specific primers will be designed for the real-time polymerase chain reaction (PCR) amplification of the genes for which the investigators have found a significant association. The miRNAs found will be analyzed after 3 months of treatment. Analysis of biomarkers. Immunoassay techniques will evaluate the following markers before and after treatment: angiotensin I, II and III, plasma renin activity, atrial natriuretic peptide (ANP), brain natriuretic peptide (BNP) and endogenous ouabain.

CONTACTS AND LOCATIONS:
Locations (1):
- Ferran Barbé, Lleida, Spain